CLINICAL TRIAL: NCT01707264
Title: A Phase 1/2, Open Label, Dose Escalation Study of Intravenous Administration of Single Agent NEOD001 in Subjects With Light Chain (AL) Amyloidosis
Brief Title: Phase 1/2, Open Label, Dose Escalation Study of NEOD001 in Subjects With Light Chain (AL) Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prothena Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEOD001-001
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Primary Amyloidosis
Keywords: AL amyloidosis; Primary amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — birtamimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NEOD001 (Experimental): NEOD001 will be administered intravenously once every 28 days. The starting dose will be 0.5 mg/kg. Dose escalation will continue until the the maximum tolerated dose is determined for single agent NEOD001. Approximately 20 additional subjects will be treated with the maximum tolerated dose.
  Interventions: Drug: NEOD001

INTERVENTIONS:
Drug: NEOD001 — Monoclonal antibody administered by intravenous infusion every 28 days.

SUMMARY:
Dose escalation study to determine the maximum tolerated dose of NEOD001 in approximately 30 subjects with AL amyloidosis. Expansion phase to evaluate safety, efficacy and pharmacokinetics of NEOD001 in 25 additional subjects at the maximum tolerated dose.

DETAILED DESCRIPTION:
The purpose of the dose escalation phase of the study is to determine the maximum tolerated dose/Phase 2 recommended dose of NEOD001 when given as a single agent intravenously in approximately 30 subjects with AL amyloidosis.

The purpose of the expansion phase of the study is to evaluate the safety, preliminary efficacy and pharmacokinetics of single agent NEOD001 at the maximum tolerated dose/Phase 2 recommended dose in approximately 25 additional evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 years;
2. ECOG performance status (PS) 0-2;
3. Diagnosis of systemic AL amyloidosis (subjects with non-AL amyloidosis are not eligible);
4. Received at least one prior systemic therapy, which may include stem cell transplant, for AL amyloidosis;
5. Have adequate organ function;
6. Ability to understand and willingness to sign informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. Secondary or familial amyloidosis;
2. Life expectancy of < 3 months;
3. Symptomatic multiple myeloma;
4. Hypersensitivities to other monoclonal antibodies;
5. Known HIV infection;
6. Women who are lactating;
7. Any other condition or prior therapy, which in the opinion of the PI, would make the subject unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-08-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 28 day cycles, up to 1 year; beyond 1 year with approval of Sponsor and Investigator
  * Adverse event profile
  * Dose limiting toxicity and maximum tolerated dose
Maximum tolerated dose | 28 day cycles, up to 1 year; beyond 1 year with approval of Sponsor and Investigator
  * Adverse event profile
  * Dose Limiting Toxicity and maximum tolerated dose

SECONDARY OUTCOMES:
Pharmacokinetics | 28 day cycles, up to 1 year; beyond 1 year with approval of Sponsor and Investigator
  • Pharmacokinetic parameters including Cmax, Tmax, AUC, Cav, Cmin, t½, CL, and Vz
Immunogenicity | 28 day cycles, up to 1 year; beyond 1 year with approval of Sponsor and Investigator
  • Measurement of anti-NEOD001 antibodies

OTHER OUTCOMES:
Hematologic Response | 28 day cycles, up to 1 year; beyond 1 year with approval of Sponsor and Investigator
  • Hematologic response
Organ response | 28 day cycles, up to 1 year; beyond 1 year with approval of Sponsor and Investigator
  * Organ response
  * Changes in organ function markers

CONTACTS AND LOCATIONS:
Overall Officials: Julia Martinisi, Study Director — Prothena Biosciences Ltd.
Locations (7):
- United States (7):
  - Stanford University Cancer Center, Palo Alto, California
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Gertz MA, Landau H, Comenzo RL, Seldin D, Weiss B, Zonder J, Merlini G, Schonland S, Walling J, Kinney GG, Koller M, Schenk DB, Guthrie SD, Liedtke M. First-in-Human Phase I/II Study of NEOD001 in Patients With Light Chain Amyloidosis and Persistent Organ Dysfunction. J Clin Oncol. 2016 Apr 1;34(10):1097-103. doi: 10.1200/JCO.2015.63.6530. Epub 2016 Feb 8. PMID 26858336